CLINICAL TRIAL: NCT04190108
Title: Frequency of Elevated Fecal Calprotectin Levels in Psoriatic Arthritis and Its Predictive Role for Inflammatory Bowel Disease Occurrence: a Prospective, Long-term, Controlled Study.
Brief Title: Frequency of Elevated Fecal Calprotectin Levels in Psoriatic Arthritis.
Status: Completed | Type: Observational
Sponsor: Hospital of Prato (Other)
Collaborators: Giulia Franchi,Department of Rheumatology, Hospital of Prato (Unknown); Maurizio Benucci,S.Giovanni di Dio Hospital (Unknown); Raffaele Scarpa, Rheumatology Unit, University of Naples Federico II, Naples (Unknown); Francesco Caso, Rheumatology Unit, University of Naples Federico II, Naples (Unknown); Rosario Foti,Rheumatology Unit, A.O.U. Policlinico Vittorio Emanuele, Catania (Unknown); Antonio Carletto,Rheumatology Unit, AOUI, Verona. (Unknown); Elisa Visalli,Rheumatology Unit, A.O.U. Policlinico Vittorio Emanuele, Catania (Unknown); Laura Niccoli,Department of Rheumatology, Hospital of Prato (Unknown)
Responsible Party: Principal Investigator, Fabrizio Cantini, MD, Hospital of Prato
Other Study IDs: HPrato-2
Record Dates: First submitted 2019-11-26; First posted 2019-12-09 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Psoriatic Arthritis; Inflammatory Bowel Diseases
MeSH Terms: conditions — Arthritis, Psoriatic; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case patients: All consecutive, new patients older than 18 years with PsA (CASPAR criteria) at onset observed over 3-year period, who had any abdominal symptoms.
  Interventions: Diagnostic Test: Fecal calprotectin assay
- Controls: All consecutive new patients meeting the ACR/EULAR 2010 classification criteria for rheumatoid arthritis (RA) at onset.
  Interventions: Diagnostic Test: Fecal calprotectin assay

INTERVENTIONS:
Diagnostic Test: Fecal calprotectin assay — FC levels were measured at baseline with Bühlmann fCAL Turbo, Switzerland® kit.

SUMMARY:
Background.Recent epidemiologic studies have shown an association between psoriasis, psoriatic arthritis (PsA) and inflammatory bowel diseases (IBD). Recently, measurement of fecal calprotectin (FC) demonstrated a good sensitivity and specificity for intestinal inflammation.

Primary objective of present study was to evaluate the presence of occult bowel inflammation in patients with PsA as expressed by elevated levels of FC. Secondary objectives were to investigate the correlation between the levels FC and clinical and laboratory features, and the outcome of CF-positive patients in terms of IBD development.

DETAILED DESCRIPTION:
A number of studies evaluated the presence of occult intestinal inflammation by using FC assay in patients with axial SpA. In 2000, a study conducted in PsA patients without bowel symptoms showed at mucosa biopsies the presence of microscopic changes, increase in lamina propria cellularity, consisting of plasma cells and lymphocytes, and lymphoid aggregates.Present prospective case-control study was designed to investigate occult intestinal inflammation by using FC assay in consecutive patients with PsA at onset, and who had no abdominal symptoms. Five Italian Centers contributed to patients recruitment adopting the same inclusion and exclusion criteria over a 3 year period.

FC levels were measured at baseline with Bühlmann fCAL Turbo, Switzerland® kit. This automated method is a particle enhanced turbidimetric immunoassay employing polyclonal antibodies. The manufacturer cut-off for FC positivity was 50 μg/g, with a sensitivity of 100% and a specificity of 53.1%.

The number of patients developing IBD was evaluated at the end of follow-up. Clinical and laboratory data collection was centralized and two experts statisticians performed the data analysis.

Statistical analysis. All demographic, clinical, and laboratory data were collected and descriptive statistics, presented as mean value and standard deviation, were calculated using Microsoft ® Office Excel for Windows and ©2019 Minitabs, LLC for Windows. Chi-square test was used for categorical variables. FC test sensitivity, specificity, positive (PPV) and negative (NPV) predictive values were calculated. Bayes's theorem was used to calculate the 95% confidence interval (95%CI). Correlations were calculated using Spearman's correlation (rs). P values ≤ 0.05 were accepted as statistically significant.

The median follow-up was 30 months.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* absence of any abdominal symptoms or diarrhoea
* non-steroidal anti-inflammatory drug (NSAIDs) interruption 10 days before enrollment
* Corticosteroids (CS) at stable low dose (prednisone 10 mg/day or equivalent) during the preceding 2 weeks were permitted in both groups.

Exclusion Criteria:

* age < 18 years
* previous diagnosis of CD or UC or current diagnosis of infectious colitis
* previous therapy with traditional DMARDs or any biologic therapies
* CS at high doses.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Both cases and controls were abdominal symptom-free.
Sampling Method: Non-Probability Sample
Enrollment: 259 (Actual)
Dates: Start 2016-01-02 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
The percentage of elevated FC levels in cases and controls | 3 YEARS
  Comparison of FC levels between cases and controls

SECONDARY OUTCOMES:
Correlations of FC levels with laboratory data | 3 YEARS
  Spearman's correlation (rs)
The percentage of patients developing IBD over the follow up | 3 YEARS
  The occurrence of IBD over the follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Fabrizio Cantini, Prato, Tuscany, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fu Y, Lee CH, Chi CC. Association of Psoriasis With Inflammatory Bowel Disease: A Systematic Review and Meta-analysis. JAMA Dermatol. 2018 Dec 1;154(12):1417-1423. doi: 10.1001/jamadermatol.2018.3631. PMID 30422277
- [Background] Scher JU, Ubeda C, Artacho A, Attur M, Isaac S, Reddy SM, Marmon S, Neimann A, Brusca S, Patel T, Manasson J, Pamer EG, Littman DR, Abramson SB. Decreased bacterial diversity characterizes the altered gut microbiota in patients with psoriatic arthritis, resembling dysbiosis in inflammatory bowel disease. Arthritis Rheumatol. 2015 Jan;67(1):128-39. doi: 10.1002/art.38892. PMID 25319745
- [Background] Klingberg E, Strid H, Stahl A, Deminger A, Carlsten H, Ohman L, Forsblad-d'Elia H. A longitudinal study of fecal calprotectin and the development of inflammatory bowel disease in ankylosing spondylitis. Arthritis Res Ther. 2017 Feb 2;19(1):21. doi: 10.1186/s13075-017-1223-2. PMID 28148281
- [Background] Adarsh MB, Dogra S, Vaiphei K, Vaishnavi C, Sinha SK, Sharma A. Evaluation of subclinical gut inflammation using faecal calprotectin levels and colonic mucosal biopsy in patients with psoriasis and psoriatic arthritis. Br J Dermatol. 2019 Aug;181(2):401-402. doi: 10.1111/bjd.17745. Epub 2019 May 6. No abstract available. PMID 30729502
- [Background] Scarpa R, Manguso F, D'Arienzo A, D'Armiento FP, Astarita C, Mazzacca G, Ayala F. Microscopic inflammatory changes in colon of patients with both active psoriasis and psoriatic arthritis without bowel symptoms. J Rheumatol. 2000 May;27(5):1241-6. PMID 10813294